CLINICAL TRIAL: NCT06163417
Title: Laparoscopic Kasai Portoenterostomy Has Similar Surgical Outcomes and Better Urine Output Compared to Standard Open Kasai- Portoenterostomy: A Ten-year Retrospective Cohort Study
Brief Title: Laparoscopic Kasai Has Similar Anesthetic Outcomes to Open Kasai
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE22128A
Record Dates: First submitted 2023-11-14; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- O group: conventional Kasai portoenterostomy
- L group: laparoscopic Kasai portoenterostomy
  Interventions: Procedure: laparoscopic

INTERVENTIONS:
Procedure: laparoscopic — laparoscopic
  Groups: L group

SUMMARY:
Biliary atresia (BA) is a rare biliary tree disease with a high incidence in eastern Asia. Kasai operation is a standard treatment for BA, and studies have shown that timely Kasai operation is crucial for better outcomes. The Kasai operation can be performed as either an open or laparoscopic technique. This study aimed to compare the differences in anesthetic management between the two surgical groups. Herein, we compared the outcomes of infants with BA who underwent the open and laparoscopic Kasai surgery.

DETAILED DESCRIPTION:
Biliary atresia is (BA) a rare biliary tree disease. This disease, which is usually found in infancy is characterized by biliary inflammation and obliteration. The incidence variate from 1 in 5000 to 20000. However, high prevalence rate up to 1 in 5-10,000 was comparatively noted in eastern Asia, especially in Japan and Taiwan. Biliary atresia can be treated by "Kasai operation" ( Kasai portoenterotomy) or liver transplantation. In the previous study, 60% of biliary atresia patients after receiving Kasai portoenterostomy could have better liver prognosis.The timing of Kasai operation is also crucial, increased age of surgery had negative influence in the long-term follow up.

Traditionally, Kasai portoenterostomy was performed by open surgery. As the progression and popularity of minimally invasive surgery, laparoscopic Kasai was first introduced in 2002 and then performed in many countries. However, the advantage of laparoscopic Kasai seems still controversial due to many indicative outcomes as early jaundice clearance, native liver survival (NLS) and liver transplantation rate within 1 year after the Kasai operation even adhesions prevention seems no better maybe worse in laparoscopic group.But in our hospital, no statistically significant differences were observed for hospital stay and outcomes (including early jaundice clearance rate, episodes of cholangitis, and 2-year native liver survival rate) between the open and the laparoscopic Kasai operations.Even the better operation view was noted in laparoscopic group but operation time seems almost all prolonged in laparoscopic one compared to open one, that makes excessive fluid infusion and hypothermia easily found in laparoscopic group . However, no hypothermia and laryngeal edema were noted in our hospital compare to previous study

ELIGIBILITY:
Inclusion Criteria:

* children who had undergone Kasai portoenterostomy between January 2011 and December 2021

Exclusion Criteria:

* severe congenital heart disease requiring surgical treatment,
* reoperation,
* a diagnosis of non-biliary atresia,
* incomplete medical records.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective cohort study was conducted at a single tertiary center in central Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
fluid intake_1 | through study completion, an average of 1 year
  intravenous fluid infusion during the operation ( ml)
fluid intake_2 | through study completion, an average of 1 year
  transfusion volume during the operation (ml)
output_1 | through study completion, an average of 1 year
  urine output
output_2 | through study completion, an average of 1 year
  blood loss (ml)

SECONDARY OUTCOMES:
respiratory outcomes_1 | through study completion, an average of 1 year
  extubation time ( duration between extubation and end of the surgery)
respiratory outcomes_2 | through study completion, an average of 1 year
  EtCO2
respiratory outcomes_3 | through study completion, an average of 1 year
  peak airway pressure
surgery duration of the surgery | through study completion, an average of 1 year
  total surgery time
total days of hospitalization | through study completion, an average of 1 year
  total hospital days
total days of admission to ICU | through study completion, an average of 1 year
  total ICU days
surgery-related outcomes_1 | through study completion, an average of 1 year
  postoperative day 1 liver function ( GOT, GPT,bilirubin in the postoperative day 1)
surgery-related outcomes_2 | through study completion, an average of 1 year
  native liver survival time ( duration before liver transplantation)
surgery-related outcomes_3 | through study completion, an average of 1 year
  cholangitis ( cholangitis needes antibiotics treatment)
surgery-related outcomes_4 | through study completion, an average of 1 year
  6-month bilirubin clearance rate ( bilirubin below standard rate at 6-month)

IPD SHARING:
Plan to Share IPD: No